CLINICAL TRIAL: NCT00877656
Title: An Open-Label Therapeutic Exploratory Clinical Trial of HuMax-CD4, a Fully Human Monoclonal Anti-CD4 Antibody, in Patients With Refractory or Relapsed Non-Cutaneous CD4+ T-Cell Lymphoma
Brief Title: HuMax-CD4 in Non-Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: ICTM, Genmab
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hx-CD4-109
Record Dates: First submitted 2009-03-25; First posted 2009-04-08 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — zanolimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CD4 (Experimental): Open label treatment arm
  Interventions: Biological: HuMax-CD4

INTERVENTIONS:
Biological: HuMax-CD4 — Active treatment

SUMMARY:
The purpose of this study is to assess the safety and efficacy of treatment of non-cutaneous T-cell lymphoma with treatment with CD4.

DETAILED DESCRIPTION:
The study is closed and all subjects have completed treatment.

The study is to evaluate the safety and efficacy of Humax CD4 with CHO vs CHO alone in subjects with non-cutaneous T cell lymphoma. The primary efficacy will be evaluated by time to relapse.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic biopsy of non cutaneous T Cell lymphoma with positive phenotype
* Relapsed or refractory to minimum of one course of chemotherapy
* Study is closed to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-08; Primary Completion 2006-01 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by survival and time to disease progression | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Abhay Patki, PhD, Study Chair — Genmab

REFERENCES:
- [Background] d'Amore F, Radford J, Relander T, Jerkeman M, Tilly H, Osterborg A, Morschhauser F, Gramatzki M, Dreyling M, Bang B, Hagberg H. Phase II trial of zanolimumab (HuMax-CD4) in relapsed or refractory non-cutaneous peripheral T cell lymphoma. Br J Haematol. 2010 Sep;150(5):565-73. doi: 10.1111/j.1365-2141.2010.08298.x. Epub 2010 Jul 14. PMID 20629661